CLINICAL TRIAL: NCT03119428
Title: A Phase 1a/b Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of OMP-313M32 Administered as a Single Agent or in Combination With Nivolumab to Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of OMP-313M32 in Subjects With Locally Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 313M32-001
Record Dates: First submitted 2017-03-29; First posted 2017-04-18 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Locally Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OMP-313M32 (Experimental): Intravenous (in the vein) infusions of OMP-313M32 as a single agent
  Interventions: Drug: OMP-313M32
- OMP-313M32 and Nivolumab (Experimental): Intravenous (in the vein) infusions of OMP-313M32 in combination with nivolumab
  Interventions: Drug: OMP-313M32; Drug: Nivolumab

INTERVENTIONS:
Drug: OMP-313M32 — OMP-313M32 is a monoclonal antibody which binds to the human TIGIT receptor on T cells.
  Other Names: Anti-TIGIT monoclonal antibody
Drug: Nivolumab — Human IgG4 anti-PD-1 monoclonal antibody
  Other Names: Opdivo
  Arms: OMP-313M32 and Nivolumab

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of OMP-31M32 as a single agent or in combination with nivolumab. OMP-313M32 is an experimental anti-TIGIT antibody that was developed to block TIGIT from binding PVR allowing the body's T-cells to destroy cancer cells.

DETAILED DESCRIPTION:
This is an open-label, Phase 1a/b dose escalation study of OMP-31M32 administered as a single agent or in combination with nivolumab to evaluate the safety, tolerability pharmacokinetics, and pharmacodynamics in patients with locally advanced or metastatic solid tumors. This study consists of a screening period, a treatment period and a post-treatment follow-up period in which patients will be followed for survival for up to 2 years. Subjects will be enrolled in two stages in the Phase 1a (dose escalation and expansion) and one stage in the Phase 1b (dose escalation).

ELIGIBILITY:
Inclusion Criteria:

1. Histologic documentation of locally advanced, recurrent or metastatic solid malignancy that has progressed and standard therapy has been ineffective or intolerable. Phase 1b subjects must also have experienced disease progression after treatment with an anti PD-1 or PDL-1 agent.
2. Ability to understand the willingness and to sign a written informed consent document
3. Age >/= 18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Life expectancy >/=12 weeks
6. Measurable disease per response evaluation criteria in solid tumors.
7. Adequate hematologic and organ function
8. For women of childbearing potential and men with partners of childbearing potential, agreement (by patient and/or partner) to use two effective forms of contraception from study entry through at least 6 months after the termination visit.

Exclusion Criteria:

1. Anti-cancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 3 weeks or 5 half lives, whichever is shorter, prior to initiation of study treatment
2. Active autoimmune disease or a history of severe autoimmune disease or syndrome
3. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
4. Inability to comply with study and follow-up procedures.
5. Pregnancy, lactation, or breastfeeding women.
6. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, or unstable angina.
7. Known clinically significant liver disease,
8. Major surgical procedure within 28 days prior to initiation of study treatment or anticipation of need for a major surgical procedure during the course of the study.
9. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | Subjects will be assessed for DLTs through the end of the first cycle (Days 1-29)
  The Maximum tolerated dose (MTD) or maximum administered dose (MAD) will be determined in patients treated with OMP-313M32 in combination with nivolumab
Incidence of treatment emergent adverse events | up to approximately 2 years
  Percentage of patients with adverse events

SECONDARY OUTCOMES:
Pharmacokinetic Outcome Measures (AUC) - Phase 1a | 1st dose and 4th dose: pre-dose, post-infusion, and 1, 3, 7 and 10 days. All other doses: pre-dose, 15 minutes and 7 days post-infusion. PK sample will be taken at treatment termination and every 4 wks for 12 wks.
  Area under the plasma concentration versus time curve (AUC) will be evaluated
Pharmacokinetic Outcome Measures (AUC) - Phase 1b | 1st dose and 4th dose: pre-dose and 15 minutes post-infusion. All other doses: pre-dose. PK sample will be taken at treatment termination and every 4 wks for 12 wks.
  Area under the plasma concentration versus time curve (AUC) will be evaluated
Pharmacokinetic Outcome Measures (T1/2) - Phase 1a | 1st dose and 4th dose: pre-dose, post-infusion, and 1, 3, 7 and 10 days. All other doses: pre-dose, 15 minutes and 7 days post-infusion. PK sample will be taken at treatment termination and every 4 wks for 12 wks.
  The half life (T1/2) of OMP-313M32 will be assessed
Pharmacokinetic Outcome Measures (T1/2) - Phase 1b | 1st dose and 4th dose: pre-dose and 15 minutes post-infusion. All other doses, pre-dose.PK sample will be taken at treatment termination and every 4 wks for 12 wks.
  The half life (T1/2) of OMP-313M32 will be assessed
Immunogenicity of OMP-313M32 | up to approximately 2 years
  Percentage of patients with anti-OMP-313M32 antibodies assessed
Objective Response | up to approximately 2 years
  Measured by Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Progression-free survival | approximately 2 years
  Measured by Response Evaluation Criteria in Solid Tumors (RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: John Lewicki, PhD, Study Director — Mereo BioPharma
Locations (5):
- United States (5):
  - Scottsdale, Scottsdale, Arizona
  - Durham, Durham, North Carolina
  - Oklahoma, Oklahoma City, Oklahoma
  - Nashville, Nashville, Tennessee
  - Salt Lake City, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mettu NB, Ulahannan SV, Bendell JC, Garrido-Laguna I, Strickler JH, Moore KN, Stagg R, Kapoun AM, Faoro L, Sharma S. A Phase 1a/b Open-Label, Dose-Escalation Study of Etigilimab Alone or in Combination with Nivolumab in Patients with Locally Advanced or Metastatic Solid Tumors. Clin Cancer Res. 2022 Mar 1;28(5):882-892. doi: 10.1158/1078-0432.CCR-21-2780. PMID 34844977